CLINICAL TRIAL: NCT00602576
Title: Randomized Phase II Study Comparing Two Schedules Of Temozolomide In Combination With Bay 43-9006 In Patients With Advanced Melanoma
Brief Title: Temozolomide and Sorafenib in Treating Patients With Metastatic or Unresectable Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000580808; 06604 (Other: Abramson Cancer Center); 802514 (Other: U Penn IRB); P30CA016520 (NIH)
Record Dates: First submitted 2008-01-25; First posted 2008-01-28 (Estimated); Results first posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage III melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Sorafenib; Temozolomide

STUDY DESIGN:
Intervention Model Description: 4 arm parallel phase II study Arms A and B are randomized to different schedules of temozolomide Arm C is prior temozolomide-refractory patients Arm D is brain metastases patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (Experimental): Patients who were temozolomide naive and had no brain metastases received oral sorafenib tosylate twice daily on days -7 to 56 of course 1 and on days 1-56 of all subsequent courses. Patients also receive oral TMZ once daily on days 1-42.
  Interventions: Drug: sorafenib tosylate; Drug: temozolomide
- Arm B (Experimental): Patients who were temozolomide naive and had no brain metastases received sorafenib tosylate as in arm A and oral TMZ once daily on days 1-5 and 29-33.
  Interventions: Drug: sorafenib tosylate; Drug: temozolomide
- Arm C (Experimental): Patient with or without treated brain metastases who were treated with prior temozolomide and progressed were treated with oral sorafenib tosylate twice daily on days -7 to 56 of course 1 and on days 1-56 of all subsequent courses. Patients also receive oral TMZ once daily on days 1-42.
  Interventions: Drug: sorafenib tosylate; Drug: temozolomide
- Arm D (Experimental): Patients with treated brain metastases were treated with sorafenib tosylate as in arm B and oral TMZ once daily on days 1-5 and 29-33.
  Interventions: Drug: sorafenib tosylate; Drug: temozolomide

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: nexavar
Drug: temozolomide — Given orally
  Other Names: temodar

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving temozolomide together with sorafenib may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying two different schedules of temozolomide when given together with sorafenib to compare how well they work in treating patients with metastatic or unresectable melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To measure the progression-free survival of patients with metastatic or unresectable melanoma with no brain metastasis or no prior treatment with temozolomide (TMZ) treated with sorafenib tosylate in combination with two different schedules (extended daily dosing vs standard dosing) of TMZ.
* To measure the progression-free survival of patients with or without brain metastasis and prior treatment with TMZ treated with sorafenib in combination with extended daily dosing of TMZ.
* To measure the progression-free survival of patients with brain metastasis and no prior treatment with TMZ treated with sorafenib in combination with standard dosing TMZ.
* To estimate the median time to progression in all patients.
* To quantify the number and percent of patients who have stable disease after 6 months of treatment (failure to progress).
* To choose the optimal combination dosing regimen for further study.

Secondary

* To estimate and define the objective response rate in these patients.
* To characterize the duration of objective responses in these patients.
* To estimate the incidence of new symptomatic brain metastasis in these patients.
* To measure overall survival of these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to prior brain metastases (yes vs no) and prior treatment with temozolomide (TMZ) (yes vs no). Patients with no prior brain metastases who did not receive prior treatment with TMZ are randomized to 1 of 2 treatment arms. These patients are further stratified according to prior treatment with sorafenib tosylate (yes vs no). Patients with or without prior brain metastases who received prior treatment with TMZ are assigned to arm I. Patients with prior brain metastases who did not receive prior treatment with TMZ are assigned to arm II.

* Arm I: Patients receive oral sorafenib tosylate twice daily on days -7 to 56 of course 1 and on days 1-56 of all subsequent courses. Patients also receive oral TMZ once daily on days 1-42.
* Arm II: Patients receive sorafenib tosylate as in arm I and oral TMZ once daily on days 1-5 and 29-33.

In both arms, courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Histologically or cytologically confirmed melanoma that is metastatic or unresectable.
2. The following groups are eligible with regard to prior therapy in either the adjuvant or metastatic disease setting:

   a) No prior therapy c) Immunotherapy consisting of Interferon, Interleukin-2 or GM-CSF. d) Chemotherapy, either single-agent or combination. Prior temozolomide is allowable e) Vaccine therapy f) Prior sorafenib is allowable

   NB: There is no limit on the number of prior therapies
3. Prior radiation therapy is allowed. However, if radiation has been administered to a lesion, there must be radiographic evidence of progression of that lesion in order for that lesion to constitute measurable disease or to be included in the measured target lesions.
4. Measurable disease by RECIST criteria. Cutaneous lesions measuring at least 1 cm will be considered. Baseline CT or MRI scans of disease sites must be performed within 4 weeks of study entry. For patients with bone metastases, a baseline bone scan must be performed within 4 weeks of study entry.
5. Age > 18 years.
6. Eastern Cooperative Oncology Group performance status of 0 or 1.
7. Baseline laboratory values (evaluated within 14 days of randomization):

   White Blood Count > 3,000/mm3 Absolute Granulocyte Count > 1,500/mm3 Platelet Count > 100,000/mm3 Serum creatinine < 2.0 x upper limit of normal (ULN) or serum creatinine clearance estimated by the MDRD formula Total Bilirubin < 1.5 x ULN (< 3.0 x ULN in the presence of Gilbert's disease AST/ALT < 2.5 x ULN (< 5.0 ULN in the presence of liver metastases) INR < 1.5 and a PTT within the upper limit of normal (if on anticoagulation baseline INR before starting anticoagulation must be <1.5)
8. Patients must have discontinued active immunotherapy (IL-2, interferon, CTLA-4, etc.) or chemotherapy at least 4 weeks prior to entering the study and recovered from adverse events due to those agents. Patients must not receive any other investigational anticancer therapy during the period on study or the four weeks prior to entry, with the exception of vaccines.
9. Patients with brain metastases must have completed radiation therapy if radiation is clinically indicated at the time of diagnosis and discontinued steroids prior to enrollment.
10. The effects of sorafenib, temozolomide on the developing human fetus are unknown. For this reason and because antiangiogenic agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant while participating in this study, she should inform her treating physician immediately. If a man impregnates a woman while participatig in this study, he should inform his treating physician immediately as well.

EXCLUSION CRITERIA

1. Patients must not have other current malignancies, other than basal cell skin cancer, squamous cell skin cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast.
2. Patients must not have a serious intercurrent illness including, but not limited to, ongoing or active infection requiring parental antibiotics, clinically significant cardiovascular disease (e.g. uncontrolled hypertension, myocardial infarction, unstable angina), New York heart association grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, or grade II or greater peripheral vascular disease within 1 year prior to study entry, or psychiatric illness/social situations that would limit compliance with study requirements.
3. Patients must not be taking cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine or phenobarbital), rifampin or St. John's wort.
4. Women must not be pregnant or breast-feeding as the agents used in this study may be teratogenic to a fetus and there is no information on the excretion of the agents or their metabolites into breast milk. All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy.
5. Because patients with immune deficiency are at increased risk of lethal infections when treated with bone marrow-suppressive therapy, HIV-positive patients are excluded from the study. For patients receiving combination anti-retroviral therapy, the potential impact of pharmacokinetic interactions with sorafenib, temozolomide is unknown. Appropriate studies may be undertaken in patients with HIV and those receiving combination anti-retroviral therapy in the future.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2008-12-21 (Actual); Study Completion 2009-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Amaravadi, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C | Arm D
Started | 38 | 40 | 38 | 53
Completed | 38 | 40 | 38 | 53
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Arm D | Total
Number analyzed (Participants) | 38 | 40 | 38 | 53 | 169
Age, Continuous [Median (Full Range); unit: years] | 62 [26 to 83] | 61 [44 to 84] | 61 [35 to 78] | 58 [37 to 83] | 61 [26 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 10 | 18 | 54
  Male | 22 | 30 | 28 | 35 | 115
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 38 | 40 | 38 | 53 | 169

OUTCOME MEASURES:

1. Primary Outcome: Rate of 6 Month Progression-Free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 38 | 40 | 38 | 53
Participants | 18 | 15 | 4 | 12

2. Secondary Outcome: Response Rate
Description: Response Rate as defined by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Approximately 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 38 | 40 | 38 | 53
Participants | 8 | 6 | 0 | 8

3. Secondary Outcome: Overall Survival Rate
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D
Number analyzed (Participants) | 38 | 40 | 38 | 53
Participants | 12 | 18 | 5 | 17

ADVERSE EVENTS:
Time Frame: 4 years
Description: the definition ofadverse event and serious adverse events were according to clinicaltrials.gov definitions
Arm/Group | Arm A | Arm B | Arm C | Arm D
Serious Adverse Events (participants affected / at risk) | 2/38 | 0/40 | 4/38 | 1/53
Other Adverse Events (participants affected / at risk) | 38/38 | 40/40 | 38/38 | 53/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=38) | Arm B (N=40) | Arm C (N=38) | Arm D (N=53)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
delayed wound healing (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CNS hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dehydration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GI perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
aterial thrombus (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=38) | Arm B (N=40) | Arm C (N=38) | Arm D (N=53)
anemia (Blood and lymphatic system disorders) | 13 (13) | 20 (20) | 9 (9) | 16 (16)
lymphopenia (Blood and lymphatic system disorders) | 30 (30) | 27 (27) | 28 (28) | 34 (34)
neutropenia (Blood and lymphatic system disorders) | 13 (13) | 6 (6) | 2 (2) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (14) | 9 (9) | 9 (9) | 17 (17)
abdominal pain (Gastrointestinal disorders) | 7 (7) | 5 (5) | 2 (2) | 6 (6)
alopecia (Skin and subcutaneous tissue disorders) | 23 (23) | 16 (16) | 5 (5) | 16 (16)
anorexia (Metabolism and nutrition disorders) | 25 (25) | 22 (22) | 18 (18) | 28 (28)
Constipation (Gastrointestinal disorders) | 21 (21) | 12 (12) | 9 (9) | 16 (16)
dehydration (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 2 (2) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 23 (23) | 19 (19) | 7 (7) | 29 (29)
Fatigue (General disorders) | 30 (30) | 29 (29) | 22 (22) | 39 (39)
Hand/foot syndrome (Skin and subcutaneous tissue disorders) | 27 (27) | 29 (29) | 17 (17) | 34 (34)
Headache (Nervous system disorders) | 7 (7) | 6 (6) | 4 (4) | 2 (2)
hoarseness (General disorders) | 6 (6) | 7 (7) | 6 (6) | 9 (9)
hypertension (Cardiac disorders) | 11 (11) | 5 (5) | 6 (6) | 14 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (13) | 10 (10) | 10 (10) | 12 (12)
Nausea (Gastrointestinal disorders) | 27 (27) | 30 (30) | 21 (21) | 31 (31)
Rash (Skin and subcutaneous tissue disorders) | 33 (33) | 34 (34) | 19 (19) | 33 (33)
stomatitis (Skin and subcutaneous tissue disorders) | 18 (18) | 15 (15) | 15 (15) | 25 (25)
Weight loss (Metabolism and nutrition disorders) | 24 (24) | 22 (22) | 14 (14) | 29 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No